CLINICAL TRIAL: NCT05498038
Title: Exercise Reset for Concussion- Modifying the Buffalo Concussion Protocol for Application in a Military Environment
Brief Title: Exercise Reset for Concussion in a Military Environment
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency); Children's Hospital of Philadelphia (Other); University of Pennsylvania (Other); University of North Carolina, Chapel Hill (Other); The Geneva Foundation (Other); Center for Neuroscience and Regenerative Medicine (CNRM) (U.S. Federal Agency); Axon Medical Technologies LLC (Industry)
Responsible Party: Principal Investigator, John J. Leddy MD, John J Leddy, MD, State University of New York at Buffalo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TP210003
Record Dates: First submitted 2022-08-09; First posted 2022-08-11 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Brain Concussion
Keywords: concussion; military; aerobic exercise; recovery; return to duty
MeSH Terms: conditions — Brain Concussion | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: This is a four-year multicenter mechanistic treatment (Phase 3) RCT that recruits CSM and healthy service members as controls. CSM who have signed a consent form to participate in the trial will be randomly assigned to either exercise+PRA or to PRA alone by the research assistant using a computer-generated randomization scheme generated by the study statistician. CSM will be allocated to trial arm using a pre-determined block randomization procedure in a 1:1 ratio, in multiples of 3 and limited to a maximum of 9, to reduce potential for imbalance across study arms. We will stratify the sample by sex and site and attempt to recruit a M:F ratio similar to the military in general (80:20). Randomization will occur without knowledge of the clinician who diagnosed the concussion. Data is collected at the first visit and weekly until clinical recovery, or up to 4 weeks from injury, and at the final 3 month time point. Controls will complete the clinic visits twice, two weeks apart.
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Healthy Control Service Members (No Intervention): Non-concussed, age-matched SM will serve as a healthy control group (HC) for comparing CSM to normal physiology and to control for the effect of time and of aerobic exercise. All HC participants will be provided with an activity monitor (with GPS tracking disabled) to wear 24 hours/day for measurement of daily physical activity and sleep duration over the time between first and final test sessions. The activity monitor also acts as an HR monitor to record the participants' HR during their prescribed exercise bouts. HC will be asked to exercise each day at approximately 70% of their age-predicted maximum heart rate (from the formula 220 minus age x 0.7 = target HR) for 20 minutes to control for the effect of exercise on the physiological tests.
- Concussed Service Members PRA (No Intervention): CSM randomized to PRA alone will receive written instructions on how to follow the PRA protocol. All participants will be provided with an activity monitor (with GPS tracking disabled), and we will record daily physical activity and sleep patterns.
- Concussed Service Members PRA+Exercise (Experimental): CSM randomized to aerobic exercise+PRA will receive their individualized aerobic exercise prescription plus written instructions on how to follow the PRA protocol. CSM will start the exercise program the day after the first visit. All participants will be reminded each day by text message to complete their assigned activity (in the case of exercise + PRA participants, to perform their exercise at the prescribed dose [HR]) and to report any adverse effects). All participants will also report symptoms once daily in response to a text message to their phone. All participants will wear an activity monitor continuously until clinical recovery or for 4 weeks to measure daily activity and sleep. The activity monitor will also act as an HR monitor and will be worn by participants in the PRA+aerobic exercise group during daily exercise sessions to measure participant adherence to the prescribed exercise dose.
  Interventions: Behavioral: Aerobic Exercise

INTERVENTIONS:
Behavioral: Aerobic Exercise — Participants are asked to complete at least 20 minutes of aerobic exercise every day, excluding clinic visits.
  Arms: Concussed Service Members PRA+Exercise

SUMMARY:
Our primary objective is to show that early, personalized aerobic exercise treatment safely improves concussion recovery, speeds RTD, and reduces persistent symptoms in CSM. Our secondary objectives include demonstrating the clinical utility of our March-in-place test and determining fundamental mechanisms for the effect of exercise rehabilitation on concussion recovery. We will conduct a prospective four-year multicenter mechanistic treatment (Phase 3) RCT in CSM of personalized sub-threshold aerobic exercise added to the PRA compared with the PRA alone. Non-concussed, age-matched SM will serve as a healthy control group (HC) for comparing CSM to normal physiology and to control for the effect of time and of aerobic exercise.

DETAILED DESCRIPTION:
Aim 1: Determine whether early sub-threshold aerobic exercise (i.e., light limited duty) added to the current Department of Defense Progressive Return to Activity [DoD PRA]) protocol speeds return to duty (RTD), improves clinical recovery, and protects against risk of persistent post-concussive symptoms (PPCS).

Hyp 1.1: Aerobic exercise+DoD PRA early after injury speeds RTD and improves clinical recovery in CSM compared to the DoD PRA protocol alone. Hyp 1.2: Early aerobic exercise+DoD PRA protects against risk of PPCS in concussed service members (CSM) at 1 and at 3 months post-injury versus the DoD PRA protocol alone.

Aim 2: Determine whether a March-in-place test informs clinical decision-making and contributes to RTD decisions. Hyp 2.1: The degree of early exercise intolerance on the Buffalo Concussion March Test (BCMT) will correlate with the development of PPCS and inform clinician decision making on RTD.

Aim 3: Determine how aerobic exercise improves concussion recovery. Hyp 3.1: Aerobic exercise improves abnormal autonomic nervous system (ANS) regulation in CSM. Hyp 3.2: Aerobic exercise improves expression of salivary brain-derived neurotrophic factor (BDNF), BDNF-related miRNAs, and inflammatory-related miRNAs seen in CSM. Hyp 3.3: Aerobic exercise improves mental health (i.e., anxiety/depressive symptoms, sleep, resilience, self-efficacy, morale) in CSM.

Aim 4: Evaluate the suitability of the Exercise RESET testing and intervention approach for military use informed by study participants and providers.

ELIGIBILITY:
Inclusion Criteria (Participants):

For the CSM Group:

* Active-duty service member
* Aged 18-40 years
* Injury occurred within 9 days of injury
* Diagnosed with concussion by an experienced clinician using standard international criteria

For the HC Group:

* Active-duty service member
* Ages 18-40

Exclusion Criteria (Participants):

For the CSM group:

* Moderate or severe TBI as indicated by a GCS score <13, lesion on CT/MRI, and/or focal neurologic sign consistent with intracerebral lesion
* Injury involving loss of consciousness for >30 minutes or post-traumatic amnesia >24 hours
* Inability to exercise because of lower-extremity orthopedic injury, clinically significant vestibular or visual dysfunction, or increased cardiac risk
* Pre-existing conditions that prevent participation in active testing and/or rehabilitation
* Active substance abuse/dependence
* Unwillingness to perform intervention
* Limited English proficiency
* Confirmed pregnancy

For the HC group:

* Has lingering symptoms from a previous concussion or has recovered from a concussion less than 1-month ago
* On a limited profile or "chit" for light duty
* Active substance abuse/dependence
* Unwilling to perform intervention
* Limited English proficiency
* Confirmed pregnancy

Inclusion Criteria (Providers):

* Active duty
* Currently active clinician (MD, DO, PT, ATC, OT) involved in concussion management beyond initial emergent diagnosis
* Willing to participate
* Able to be contacted by telephone or Zoom

Exclusion Criteria (Providers):

* Not active duty
* Not currently an active clinician (MD, DO, PT, ATC, OT) involved in concussion management
* Only involved in concussion management at emergent timepoint
* Unwilling to participate
* Unable to be contacted by telephone or Zoom

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 168 (Estimated)
Dates: Start 2024-08-07 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Persistent Post Concussive Symptoms (PPCS) (Yes/No) | 28 days
  PPCS is defined as recovery more than 28 days from the day of concussive injury (yes) or before 28 days (no). Recovery is defined as return to baseline symptoms, exercise tolerant and confirmation by independent medical examination.
Days until Recovery | 3 months
  Determination of clinical recovery will be made by a clinician. Each week we will use a multi-modal assessment to establish clinical recovery, which is defined as return to a pre-injury level of symptoms, a normal physical examination and exercise tolerant on the graded exercise assessment.
Neurobehaviorial Symptom Inventory-22 (NSI) | 4 years
  To assess ongoing concussion symptoms, one of the main outcomes of the study. The NSI is a 5-minute measure validated in military populations to characterize concussion symptoms, endorsed by VA/DoD as a core TBI outcome measure. We will also use the symptom scale of the NSI to ask CSM about symptoms that existed before the concussion.
Average weekly Physical Activity time | 4 years
  Average of activity time per day over one week (hours:minutes) - Physical activity is measured using Polar Coach to control for this potential mediator of concussion recovery. Activity time in duration per day (hours:minutes) is tracked and then manually averaged and recorded via a standardized Excel spreadsheet.
Buffalo Concussion March-in-place Test (BCMT) | 4 years
  Average total steps per day over one week- Physical activity is measured using Polar Coach to control for this potential mediator of concussion recovery. Total steps per day are tracked and then manually averaged and recorded via a standardized Excel spreadsheet.
Daily Symptom Score Severity | 4 years
  Daily Symptom Score Severity will be measured using Ecological Momentary Assessment (EMA) (RECOUPS) - Measure daily symptoms to control for this potential mediator of concussion recovery. Participants report their symptom score once daily in response to text messages sent to their smartphone.
Average Nightly Sleep Quality | 4 years
  Measure sleep quality using Polar Coach to control for this potential mediator of concussion recovery. Duration of sleep time, sleep start time, sleep end time, and sleep restlessness score of each sleep session are tracked. Average sleep time per night, average sleep continuity, and average sleep continuity percentages are recorded via a standardized Excel spreadsheet and summated to generate a sleep quality score which will be analzyed.

SECONDARY OUTCOMES:
Concentration of Salivary BDNF | 4 years
  Concentration of salivary BDNF will be collected and used as a measure to assess enhanced neuroplasticity as a possible mechanism for the effect of aerobic exercise treatment on concussion.
Salivary miRNA | 4 years
  Concentration of salivary miRNA will be collected and used as a measure to assess enhanced neuroplasticity as a possible mechanism for the effect of aerobic exercise treatment on concussion.
National Institute of Neurological Disorders Scale (NIHSS) | 4 years
  We will collect brief validated measures of anxiety and depression to assess improved mental health as a potential mechanism for the effect of aerobic exercise treatment on concussion. Low scores indicate no deficit in neurological symptoms; high scores indicate severe deficits in neurological symptoms, and values range from 0 to 42.
Stroke Patient Reported Outcomes and Measurement Information System (PROMIS) scale | 4 years
  We will collect brief validated measures of anxiety and depression to assess improved mental health as a potential mechanism for the effect of aerobic exercise treatment on concussion. Higher scores compared to the general population via standardized T-Scores indicate impairments, and values range from 20 to 80.
The Health Care Climate Questionnaire (HCCQ) | 4 years
  We will collect brief validated health care related measures that follow Self - Determination Theory. The HCCQ measures the degree an individual feels autonomy-supported or controlled within the healthcare context, with higher scores indicating more autonomy and support felt. The range of scores is 15 to 105.
PTSD- Military Checklist (PCL-M) | 4 years
  We will collect brief validated health care related measures that follow Self - Determination Theory. The PCL-M measures the degree an individual exhibits PTSD symptoms, with higher scores indicating higher likelihood of PTSD. The range of scores is from 17 to 85.
Brief Resilience Survey (BRS) | 4 years
  We will measure resilience using this scale, which has been used to evaluate the effect on concussion recovery after sport- related concussion. Higher scores indicate more resilience, and scores range from 6 to 30.
Army Command Climate Survey | 4 years
  We will use this scale to measure morale. Higher scores indicate higher feelings of morale in units, and scores range from 2 to 10.
Cervical Range of Motion | 4 years
  Cervical Range of Motion (ROM) in degrees will be measured using the NeckCare device, an electronic medical device worn on the head to provide reliable assessments. Range of values is based on individual ability, with lower values indicating less ROM and higher values indicating more ROM.
Joint Position Error (JPE) | 4 years
  Joint Position Error (JPE) in degrees will be measured using the NeckCare device, an electronic medical device worn on the head to provide reliable assessments. Range of values is based on individual ability, with lower values indicating more precise proprioceptive capabilities, and higher values indicating less precise proprioceptive capabilities.
The Butterfly Test | 4 years
  Movement sense and eye-head-neck coordination using a score to control values will be measured using the NeckCare device, an electronic medical device work on the head to provide reliable assessments. Range of values is based on individual abilities compared to standard values, with lower values indicating more precise proprioceptive capabilities, and higher values indicating less precise proprioceptive capabilities.
Heart Rate Variability (HRV) milliseconds | 4 years
  HRV, measured as R-R intervals in ms, will be measured using the Elite HRV app 5 minutes pre-post exercise. This will be used to assess parasympathetic autonomic function as a possible mechanism for the beneficial effect of aerobic exercise treatment.
The rate of HR recovery after the BCMT in beats per minute (BPM) | 4 years
  The difference in HR from the immediate cessation of exercise to two minutes post-exercise will be used to assess parasympathetic autonomic function as a possible mechanism for the beneficial effect of aerobic exercise treatment.
Pupillary reaction time | 4 years
  Pupillary reaction (time in milliseconds) will be assessed using the Intellig-eyes system. This will be used to assess parasympathetic autonomic function as a possible mechanism for the beneficial effect of aerobic exercise treatment.
Pupil diameter change | 4 years
  Pupil diameter change will be measured in mm assessed using the Intellig-eyes system. This will be used to assess parasympathetic autonomic function as a possible mechanism for the beneficial effect of aerobic exercise treatment.
Convergence rate millseconds | 4 years
  Convergence rate (in ms) will be assessed using the Intellig-eyes system. This will be used to assess parasympathetic autonomic function as a possible mechanism for the beneficial effect of aerobic exercise treatment.
Time of Completion wioth the King Devick (KD) pre and post-exercise | 4 years
  We will use the KD test to assess for exercise-induced vision dysfunction (EIVD). Higher time (in seconds) indicates more dysfucntion indicative of concussion.
Number of errors on the King Devick (KD) pre and post-exercise | 4 years
  We will use the KD test to assess for exercise-induced vision dysfunction (EIVD). Higher number of errors indicates more dysfunction indicative of concussion.
Run/roll/aim task | 4 years
  We will use the run/roll/aim task to assess symptom change pre and post high demand vestibular activity.
Suitability of Exercise RESET | 4 years
  Study participants who complete test procedures will be invited to participate in a semi-structured interview with the intention to learn about how the intervention worked or did not work for and to get feedback about how the intervention might be improved for implementation in a military environment. On site providers who engage in concussion care will also be invited for a separate semi-structured interview to provide insights on the acceptability of the Buffalo Protocol in the military health care setting.

CONTACTS AND LOCATIONS:
Overall Officials: John Leddy, MD, Principal Investigator — University at Buffalo
Locations (2):
- United States (2):
  - Fort Liberty, Fayetteville, North Carolina
  - Camp LeJeune, Jacksonville, North Carolina

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared.